CLINICAL TRIAL: NCT04822363
Title: The Accuracy Of A Novel Platelet Activity Assay In Humans On Antiplatelet Agents: Pharmacodynamics And Comparison With Light Transmission Aggregometry
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Rushad Patell, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-P-000134
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Platelet Activation Testing Before/After Anti-platelet Therapy; Healthy
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A: Healthy (Experimental): Low Dose Aspirin - 81mg daily for 7 days
  Interventions: Drug: Aspirin
- Group B: Healthy (Experimental): High Dose Aspirin - 325mg daily for 7 days
  Interventions: Drug: Aspirin
- Group C: Healthy (Experimental): Clopidogrel 300mg on Day 1 and 75mg daily for 6 subsequent days
  Interventions: Drug: Clopidogrel
- Group D: Obese (Experimental): Low Dose Aspirin - 81mg daily for 7 days
  Interventions: Drug: Aspirin
- Group E: Obese (Experimental): Clopidogrel 300mg on Day 1 and 75mg daily for 6 subsequent days
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — Low dose aspirin in Arms A and D and High Dose Aspirin in Arm B
  Arms: Group A: Healthy; Group B: Healthy; Group D: Obese
Drug: Clopidogrel — Arms C and E
  Arms: Group C: Healthy; Group E: Obese

SUMMARY:
The purpose of this study is to test a novel diagnostic immunoassay of platelet function and compare it to the current gold standard platelet function assay by testing the response to aspirin and clopidogrel in a group of healthy volunteers and severely obese individuals and comparing the accuracy of the two tests. The secondary goals will be to evaluate the pharmacodynamic parameters of the antiplatelet agents across the two testing modalities and refine the cutoffs used for the novel assay.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subject is willing to participate and provide informed consent
3. Subject is considered reliable and capable of adhering to the protocol per the judgment of the Investigator
4. Groups A, B and C: BMI < 30 kg/m2; Groups D and E: BMI ≥ 35 kg/m2
5. Subjects must be age ≥ 18 years old
6. Serum Creatinine < 1.5 mg/dL
7. Platelet count ≥ 150 K/uL
8. Hematocrit ≥ 38%

Exclusion Criteria:

1. Pregnant. If female of child-bearing age, negative urinary pregnancy test required at time of enrollment. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant she should inform her treating physician immediately.
2. Established diagnosis of cirrhosis or active cancer
3. History of allergy to aspirin or clopidogrel
4. Any history of taking aspirin, antiplatelet drugs, NSAIDS, cyclooxygenase (COX)-2 inhibitors, warfarin, low-molecular weight heparin, thrombolytic agents, or other anticoagulants (such as direct thrombin inhibitors or factor X inhibitors) within 2 weeks prior to enrollment. (Refer to appendix)
5. Use of certain antibiotics, cardiovascular drugs, lipid-lowering agents, antidepressants, antihistamines, non-prescription drugs, and supplements within the past 2 weeks. (Refer to appendix)
6. Any major illness requiring hospitalization or surgery in the previous six months.
7. Personal history of gastrointestinal bleed in the last 24 months or diagnosis of peptic ulcer disease in the last 12 months
8. Lifetime personal history of hemorrhagic stroke.
9. Personal or family history of bleeding diatheses, including hemophilias, von Willebrand's disease, Bernard-Soulier syndrome, or Glanzmann thrombasthenia (unless otherwise confirmed not present in study subject)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison at day 5 of pDrp1 Assay relative to Light Transmission Aggregometry | 5 days
  Sensitivity of pDrp1 assay for platelet inhibition at day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided